CLINICAL TRIAL: NCT03024359
Title: Effect of Monounsaturated Fatty Acids Consumption in Brown/Beige Adipose Tissue Activity in Human Adults
Brief Title: Monounsaturated Fatty Acids and Brown/Beige Adipose Tissue in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Milena Monfort Pires, LDN, MSc, PhD, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CAAE: 60698716.1.0000.5404
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Obese
Keywords: Obesity; Brown adipose tissue; Monounsaturated fatty acids; Hypothalamic inflammation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: All subjects receive a dietary intervention with olive oil.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- obese individuals (Active Comparator): Individuals with BMI between 30 and 35 kg/m2 will be included in this group and will receive 4 weeks of extra virgin olive oil. Before and after the intervention period data regarding dietary intake and physical activity, brown/beige adipose tissue activity, body composition (DXA), lipid profile and inflammatory markers and brain activity (18F-FDG PET/MRI; in a subsample of 5 obese individuals)will be collected.
  Interventions: Dietary Supplement: Extra virgin olive oil
- normal weight individuals (Active Comparator): Individuals with BMI between 18.5 and 24.99 kg/m2 will be included in this group and will receive 4 weeks of extra virgin olive oil. Before and after the intervention period data regarding dietary intake and physical activity, brown/beige adipose tissue activity, body composition (DXA), lipid profile and inflammatory markers and and brain activity (18F-FDG PET/MRI; in a subsample of 10 normal weight individuals) will be collected.
  Interventions: Dietary Supplement: Extra virgin olive oil

INTERVENTIONS:
Dietary Supplement: Extra virgin olive oil — 2 liters of extra virgin olive oil will be given to participants to include/use in their daily foods.

SUMMARY:
Considering the high prevalence of obesity its comorbidities in Brazil and in the world, different therapeutic measures have been suggested. It is currently known that brown/beige adipose tissue plays an important role in body weight control and there is strong evidence that its activity is inversely associated with obesity and metabolic diseases. Recent studies have shown an important role foods and nutrients in the activation of brown/beige adipose tissue, almost exclusively in animal models. The benefits of monounsaturated fatty acids to metabolism have been described in several studies, however, the effects of consuming large amounts of olive oil in the activity of brown/beige adipose tissue in humans have not been explored. The aim of the study is to evaluate the impact of the consumption of large amounts of extra virgin olive oil in the activity of brown/beige adipose tissue in lean and obese humans. This will be a clinical trial with a total duration of 4 weeks. Obese and controls (normal weight) participants will undergo a dietary intervention for 4 weeks with extra virgin olive oil. Before and after the intervention period several data will be collected: dietary intake and physical activity data, evaluation of brown/beige adipose tissue (with 18F-fluorodeoxyglucose positron emission tomography and magnetic resonance imaging - PET/RMI), assessment of body composition (DXA), lipid profile and inflammatory markers as well as hypothalamic inflammation (functional magnetic resonance imaging) and brown adipose tissue biopsies in a subsample of 20 participants. The data will be expressed as mean and standard deviation and the variables compared by the Student t test or ANOVA for repeated measures.

DETAILED DESCRIPTION:
1. HYPOTHESIS The effects of fatty acids consumption on brown / beige adipose tissue have not yet been explored in humans. However, studies that evaluated the effects of saturated fatty acid replacement by monounsaturated fatty acids (MUFAs) or polyunsaturated fatty acids (PUFAs) on animal and human models have observed an improvement in cardiovascular risk factors, such as reduction of subclinical inflammation, improvement of lipid profile and increase in insulin sensitivity. The mechanisms by which these fatty acids act in the improvement of risk factors have not been completely clarified and it is possible that there is an association between the reduction of cardiovascular risk factors and the activation of brown / beige adipose tissue.

   Our hypothesis is that consuming extra virgin olive oil in high amounts for one month will promote increased brown adipose tissue (BAT) activity of the participants and improve the cardiovascular risk profile, as assessed by inflammatory markers. It is possible that the response of lean and obese subjects to dietary intervention is different and that the behavior of BAT is not equal in both groups.
2. OBJECTIVE To evaluate the impact of the consumption of large amounts of extra virgin olive oil (source of monounsaturated fatty acids) on the activity of brown / beige adipose tissue in lean and obese humans.

   2.1 Specific objectives • To investigate the activity of brown and beige adipose tissue by FDG PET / RMI, before and after four weeks of intervention with high amount of extra virgin olive oil; • To evaluate the expression of BAT activity markers: uncoupling protein 1 (UCP-1), PR domain containing 16 (PRDM16), Peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α), iodothyronine deiodinase 2 (Dio2) in mononuclear cells in the whole sample;
   * To evaluate levels of fatty acids in the blood by gas chromatography, before and after the intervention to evaluate changes in fatty acid intake;
   * To evaluate concentrations of pro and anti-inflammatory cytokines in the blood before and after 4 weeks of intervention: tumor necrosis factor alpha (TNF-α), interleukin 1-beta (IL1β), Monocyte Chemoattractant Protein-1 (MCP-1), interleukin-6 and interleukin-10);
   * To evaluate the effects of interventions on metabolic markers before and after the intervention: leptin, insulin, glucose, total cholesterol and fractions, triglycerides;
   * To evaluate the effects of the intervention on anthropometry (weight, abdominal circumference) and on the body composition evaluated by Dual-energy X-ray absorptiometry (DXA);
   * To evaluate the effects of dietary interventions on brain activity (by PET/MRi) in a subsample of 15 individuals.
3. MATERIALS AND METHODS This will be an open clinical trial lasting for four weeks. The study consists of two data collections before and after a 4-week dietary intervention in which participants will be required to consume extra-virgin olive oil provided by the researchers.

   The collection of socio demographic, dietary and physical activity data, as well as the PET / MRI and the blood collections of 50 participants will be carried out at the Nuclear Medicine Center of the Medical School of the University of São Paulo. Bone densitometry (DXA) will be performed at the School of Public Health of the University of São Paulo.

   Selection of participants:

   The estimated number of individuals with a detectable brown adipose tissue (50) is 50%, with the proportion of individuals with detectable brown adipose tissue. It will include 15 obese individuals (degree I obesity) and 35 control subjects (normal weight individuals). Participants will be selected through print and electronic media.

   • Inclusion criteria For the group with obesity: Both genders, age between 25 and 40 years, BMI ≥ 30 and <35 kg / m2.

   For the normal weight group (control): Both genders, age between 25 and 40 years, BMI <25 kg / m2.
   * Exclusion Criteria

     1) Residing outside of São Paulo / Campinas; 2) pregnant women; 3) patients with severe or non-stabilized neurological or psychiatric problems; 4) use of anti-obesity or lipid-lowering medication; 5) use of adrenergic or benzodiazepine drugs; 6) individuals with neoplasms, transmissible and rheumatic diseases, hepatic or renal insufficiency, untreated thyroid dysfunction; Diabetes mellitus; 7) change of more than 5% of body weight in the last six months; 8) to be carrying out some kind of diet or modification in the usual dietary pattern; 9) have metal prostheses.
   * Design This is an open clinical trial with a total duration of four weeks. Obese and controls participants will be enrolled into a dietary intervention for 4 weeks with extra virgin olive oil (MUFA rich). Extra-virgin olive oil (2 liters) is provided to participants and the researchers adivice the participants to use the oil in all preparations during the four weeks.

   Before and after each intervention period the following data will be collected:

   - Food consumption: 24-hour recall (before and after dietary intervention) and 3-day food diary;
   * Physical activity data: International Physical Activity Questionnaire (IPAQ);
   * Evaluation of brown / beige adipose tissue volume and activity:

   Positron emission tomography with fluoride-18-labeled fluorodeoxyglucose (18F-FDG) in combination with magnetic resonance (PET / MRi).

   For the FDG PET / RMI the participants will be allocated in a room with controlled temperature (19 degrees), with light clothes and a cooling vest for 2 hours.

   - Body composition assessment: Weight (digital scale) and height (fixed stadiometer);; abdominal circumference; body composition: by Dual-energy X-ray absorptiometry (DXA);

   - Biochemical dosages: plasma glucose, triglycerides, total cholesterol and HDL-c will be determined routinely and inflammatory markers will be determined by enzyme-linked immunosorbent assay (ELISA);

   - Expression of UCP-1, PGC-1α, PRDM16 and Dio2 will be performed by Real-Time Polymerase chain reaction (RT-PCR);

   - Composition of fatty acids in plasma will be determined by gas chromatography;

   - Brain activity: will be performed in a subsample of 15 individuals using 18F-FDG PET/MRi.

   • Statistical analysis Data will be expressed as mean and standard deviation and the variables compared by Student's t-test or ANOVA for repeated measures.

ELIGIBILITY:
Gender: Both Age: 25 to 40 years

Body mass index (BMI):

Normal body weight group: BMI lower than 25 kg/m2 Obese group: BMI between 30 and 35 kg/m2

Exclusion Criteria:

1. Living outside of São Paulo;
2. pregnant women;
3. patients with severe or non-stabilized neurological or psychiatric problems;
4. use of anti-obesity or lipid-lowering medication;
5. use of adrenergic or benzodiazepine drugs;
6. individuals with neoplasms, transmissible and rheumatic diseases, hepatic or renal insufficiency, untreated thyroid dysfunction; Diabetes mellitus;
7. individuals that changed more than 5% of body weight in the last six months; 8) to be carrying out some kind of diet or modification in the usual dietary pattern; 9) having metal prostheses.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Brown adipose tissue activity measured by increase in mean standardized disposal value (SUV) | Four weeks
  We will investigate whether 4 weeks of olive oil consumption can increase the activity of brown adipose tissue measured by mean standardized disposal value (volume) using magnetic resonance imaging

SECONDARY OUTCOMES:
Hypothalamic inflammation | Four weeks
  To see whether the consumption of 4 weeks of olive oil is able to reduce hypothalamic inflammation in lean and obese individuals as measured by functional resonance imaging
Lipid profile | Four weeks
  To see whether the consumption of 4 weeks of olive oil is able to reduce LDL and total cholesterol, as well as triglycerides concentrations
Inflammatory markers | Four weeks
  To see whether the consumption of 4 weeks of olive oil is able to reduce pro-inflammatory markers (TNF-alpha, interleukin-1beta) and increase interleukin-10

CONTACTS AND LOCATIONS:
Overall Officials: Milena Monfort-Pires, PhD, Principal Investigator — University of Campinas; Licio A Velloso, Professor, Study Director — University of Campinas
Locations (1):
- Faculdade de Ciências Médicas Unicamp, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Marken Lichtenbelt WD, Vanhommerig JW, Smulders NM, Drossaerts JM, Kemerink GJ, Bouvy ND, Schrauwen P, Teule GJ. Cold-activated brown adipose tissue in healthy men. N Engl J Med. 2009 Apr 9;360(15):1500-8. doi: 10.1056/NEJMoa0808718. PMID 19357405
- [Background] Vijgen GH, Bouvy ND, Teule GJ, Brans B, Hoeks J, Schrauwen P, van Marken Lichtenbelt WD. Increase in brown adipose tissue activity after weight loss in morbidly obese subjects. J Clin Endocrinol Metab. 2012 Jul;97(7):E1229-33. doi: 10.1210/jc.2012-1289. Epub 2012 Apr 24. PMID 22535970
- [Background] Chondronikola M, Annamalai P, Chao T, Porter C, Saraf MK, Cesani F, Sidossis LS. A percutaneous needle biopsy technique for sampling the supraclavicular brown adipose tissue depot of humans. Int J Obes (Lond). 2015 Oct;39(10):1561-4. doi: 10.1038/ijo.2015.76. Epub 2015 Apr 29. PMID 25920777
- [Derived] Monfort-Pires M, U-Din M, Nogueira GA, de Almeida-Faria J, Sidarta-Oliveira D, Sant'Ana MR, De Lima-Junior JC, Cintra DE, de Souza HP, Ferreira SRG, Sapienza MT, Virtanen KA, Velloso LA. Short Dietary Intervention with Olive Oil Increases Brown Adipose Tissue Activity in Lean but not Overweight Subjects. J Clin Endocrinol Metab. 2021 Jan 23;106(2):472-484. doi: 10.1210/clinem/dgaa824. PMID 33180910